CLINICAL TRIAL: NCT05064059
Title: A Phase 3 Study of MK-4280A (Coformulated Favezelimab [MK-4280] Plus Pembrolizumab [MK-3475]) Versus Standard of Care in Previously Treated Metastatic PD-L1 Positive Colorectal Cancer (KEYFORM-007)
Brief Title: A Study of Coformulated Favezelimab/Pembrolizumab (MK-4280A) Versus Standard of Care in Subjects With Previously Treated Metastatic PD-L1 Positive Colorectal Cancer (MK-4280A-007)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4280A-007; MK-4280A-007 (Other: MSD); jRCT2031210482 (Registry Identifier: jRCT(Japan Registry of Clinical Trials)); 2024-511043-25-00 (Registry Identifier: EU CT); U1111-1302-9933 (Registry Identifier: UTN); 2021-001309-60 (EudraCT Number)
Record Dates: First submitted 2021-09-29; First posted 2021-10-01 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1),; Programmed Cell Death Receptor Ligand 1 (PDL1, PD-L1); Programmed Cell Death Receptor Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Colorectal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; regorafenib; trifluridine tipiracil drug combination

STUDY DESIGN:
Masking Description: None (Open-label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Favezelimab/Pembrolizumab (Experimental): Participants will receive coformulated favezelimab/pembrolizumab (800 mg/200 mg) intravenously (IV) on Day 1, then every 3 weeks (Q3W), for up to 35 infusions.
  Interventions: Biological: favezelimab/pembrolizumab
- Standard of Care (Regorafenib or TAS-102) (Active Comparator): At the Investigator's choice, participants will receive 160 mg regorafenib orally daily on Days 1-12 of each 28-day cycle or 35 mg/m^2 TAS-102 orally twice daily on Days 1-5 and Days 8-12 of each 28-day cycle.
  Interventions: Drug: regorafenib; Drug: TAS-102

INTERVENTIONS:
Biological: favezelimab/pembrolizumab — Coformulated favezelimab/pembrolizumab (800 mg/200 mg), IV infusion
  Other Names: MK-4280A
  Arms: Favezelimab/Pembrolizumab
Drug: regorafenib — Oral
  Other Names: STIVARGA®; REGONIX®
  Arms: Standard of Care (Regorafenib or TAS-102)
Drug: TAS-102 — Oral
  Other Names: LONSURF®
  Arms: Standard of Care (Regorafenib or TAS-102)

SUMMARY:
The purpose of this study is to assess the safety and efficacy of coformulated favezelimab/pembrolizumab (MK-4280A) in participants with metastatic colorectal cancer. The study will also compare MK-4280A with the standard of care treatment of regorafenib and TAS-102 (trifluridine and tipiracil).

The primary study hypothesis is that coformulated favezelimab/pembrolizumab (MK-4280A) is superior to standard of care with respect to overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed colorectal adenocarcinoma that is metastatic and unresectable.
* Has measurable disease per RECIST 1.1 as assessed by the local site investigator.
* Has been previously treated for the disease and radiographically progressed on or after or could not tolerate standard treatment.
* Submits an archival (≤ 5 years) or newly obtained tumor tissue sample or newly obtained tumor tissue sample that has not been previously irradiated.
* Has an Eastern Cooperative Oncology Group Performance Score (ECOG PS) of 0 to 1 within 10 days prior to first dose of study intervention.
* Has a life expectancy of at least 3 months, based on the investigator assessment.
* Has the ability to swallow and retain oral medication and not have any clinically significant gastrointestinal abnormalities that might alter absorption.
* Has adequate organ function.

Exclusion Criteria:

* Has previously been found to have deficient mismatch repair/microsatellite instability-high (dMMR/MSI-H) tumor status.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis or leptomeningeal disease.
* Has a history of acute or chronic pancreatitis.
* Has neuromuscular disorders associated with an elevated creatine kinase (eg, inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.
* Has urine protein greater than or equal to 1g/24h.
* A woman of childbearing potential who has a positive urine/serum pregnancy test within 24/72 hours prior to the first dose of study intervention.
* Has received prior therapy with an anti-programmed cell death 1 (PD-1), anti-programmed death ligand 1 (PD-L1), or anti-programmed cell death ligand 2 (PD-L2), anti-lymphocyte activation gene 3 (LAG-3) antibody, with a tyrosine kinase inhibitor (TKI; eg, lenvatinib) other than rapidly accelerated fibrosarcoma (RAF) inhibitors (binimetinib is permitted if combined with a RAF inhibitor), or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4, OX-40, cluster of differentiation [CD] 137).
* Has previously received regorafenib or TAS-102.
* Has received prior systemic anticancer therapy including investigational agents within 28 days before randomization.
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy (eg, tuberculosis, known viral or bacterial infections, etc.).
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has known history of Hepatitis B or known active Hepatitis C virus infection.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (152):
- United States (15):
  - Georgetown University Hospital ( Site 1148), Washington D.C., District of Columbia
  - Sibley Memorial Hospital ( Site 1143), Washington D.C., District of Columbia
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital-Research ( Site 1118), Marietta, Georgia
  - Norton Cancer Institute ( Site 1139), Louisville, Kentucky
  - Rutgers Cancer Institute of New Jersey ( Site 1105), New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center ( Site 1703), New York, New York
  - Oregon Health & Science University ( Site 1141), Portland, Oregon
  - MUSC Hollings Cancer Center ( Site 1715), Charleston, South Carolina
  - The West Clinic, PLLC dba West Cancer Center ( Site 1149), Germantown, Tennessee
  - UT Southwestern Medical Center ( Site 1709), Dallas, Texas
  - Intermountain Medical Center ( Site 1707), Murray, Utah
  - Inova Schar Cancer Institute ( Site 1130), Fairfax, Virginia
  - VCU Health Adult Outpatient Pavillion ( Site 1712), Richmond, Virginia
  - Blue Ridge Cancer Care ( Site 1718), Roanoke, Virginia
  - Seattle Cancer Care Alliance ( Site 1107), Seattle, Washington
- Australia (6):
  - Westmead Hospital ( Site 0057), Westmead, New South Wales
  - Royal Brisbane and Women s Hospital ( Site 0058), Herston, Queensland
  - Queen Elizabeth Hospital ( Site 0050), Woodville South, South Australia
  - Frankston Hospital ( Site 0056), Frankston, Victoria
  - Western Health-Sunshine & Footscray Hospitals ( Site 0052), St Albans, Victoria
  - St John of God Subiaco Hospital ( Site 0051), Perth, Western Australia
- Canada (3):
  - London Regional Cancer Program - London HSC ( Site 0154), London, Ontario
  - The Ottawa Hospital ( Site 0151), Ottawa, Ontario
  - Princess Margaret Cancer Centre-Division of Medical Oncology and Hematology ( Site 0155), Toronto, Ontario
- Chile (8):
  - IC La Serena Research ( Site 0202), La Serena, Coquimbo Region
  - Clinica Puerto Montt ( Site 0211), Port Montt, Los Lagos Region
  - Fundacion Arturo Lopez Perez FALP ( Site 0208), Santiago, Region M. de Santiago
  - Oncovida ( Site 0209), Santiago, Region M. de Santiago
  - Clínica Vespucio ( Site 0205), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0206), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0200), Santiago, Region M. de Santiago
  - Centro Investigacion Cancer James Lind ( Site 0204), Temuco, Región de la Araucanía
- China (24):
  - The Second Affiliated Hospital of Anhui Medical University ( Site 1179), Hefei, Anhui
  - Chongqing Cancer Hospital ( Site 1151), Chongqing, Chongqing Municipality
  - Fujian Province Cancer Hospital ( Site 1178), Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center ( Site 1150), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 1154), Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University ( Site 1159), Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 1158), Nanning, Guangxi
  - Hainan General Hospital ( Site 1177), Haikou, Hainan
  - Wuhan Union Hospital Cancer Center ( Site 1162), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 1152), Wuhan, Hubei
  - Xiangya Hospital Central South University ( Site 1171), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 1174), Changsha, Hunan
  - The Third Xiangya Hospital of Central South University ( Site 1175), Changsha, Hunan
  - Changzhou Cancer Hospital-Department of Oncology ( Site 1183), Changzhou, Jiangsu
  - Affiliated Hospital of Jiangnan University(Wuxi Fourth People's Hospital ) ( Site 1185), Wuxi, Jiangsu
  - Jilin Cancer Hospital ( Site 1163), Changchun, Jilin
  - Jinan Central Hospital ( Site 1167), Jinan, Shandong
  - Shanghai Tenth People's Hospital ( Site 1170), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center ( Site 1176), Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University ( Site 1172), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital ( Site 1161), Tianjin, Tianjin Municipality
  - Yunnan Province Cancer Hospital-Colorectal surgery ( Site 1169), Kunming, Yunnan
  - Zhejiang Cancer Hospital ( Site 1180), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital-Medical Oncology ( Site 1173), Hangzhou, Zhejiang
- Czechia (7):
  - Masarykuv onkologicky ustav ( Site 1203), Brno, Brno-mesto
  - Fakultni nemocnice v Motole ( Site 1201), Prague, Praha, Hlavni Mesto
  - Fakultni nemocnice Hradec Kralove ( Site 1207), Hradec Králové
  - Fakultni nemocnice Olomouc ( Site 1204), Olomouc
  - Fakultni nemocnice Kralovske Vinohrady ( Site 1208), Prague
  - Fakultni Thomayerova nemocnice ( Site 1205), Prague
  - Fakultni nemocnice Na Bulovce ( Site 1202), Prague
- France (5):
  - CHU Bordeaux Haut-Leveque ( Site 0305), Pessac, Gironde
  - CHU Hotel Dieu Nantes ( Site 0303), Nantes, Pays de la Loire Region
  - Institut du Cancer Avignon-Provence ( Site 0306), Avignon, Vaucluse
  - CHU Poitiers ( Site 0304), Poitiers, Vienne
  - Hopital Europeen Georges Pompidou ( Site 0300), Paris
- Germany (7):
  - LMU Klinikum Grosshadern der Universitaet Muenchen ( Site 1253), Munich, Bavaria
  - Philipps-Universitaet Marburg. ( Site 1252), Marburg, Hesse
  - Klinikum Wolfsburg ( Site 1256), Wolfsburg, Lower Saxony
  - Johanniter Krankenhaus Bonn ( Site 1254), Bonn, North Rhine-Westphalia
  - Kliniken Maria Hilf GmbH ( Site 1255), Mönchengladbach, North Rhine-Westphalia
  - Universitätsklinikum Halle ( Site 1251), Halle, Saxony-Anhalt
  - Katholisches Marienkrankenhaus gGmbH ( Site 1257), Hamburg
- Israel (7):
  - Assuta Ashdod Public ( Site 0507), Ashdod
  - Rambam Health Care Campus-Oncology Division ( Site 0500), Haifa
  - Bnei Zion Medical Center ( Site 0506), Haifa
  - Hadassa Ein Karem Medical Center ( Site 0504), Jerusalem
  - Rabin Medical Center ( Site 0503), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0501), Ramat Gan
  - Sourasky Medical Center ( Site 0502), Tel Aviv
- Italy (6):
  - Policlinico Gemelli di Roma ( Site 0552), Roma, Abruzzo
  - IRCCS Casa Sollievo della Sofferenza ( Site 0554), San Giovanni Rotondo, Foggia
  - Istituto Clinico Humanitas - Cancer Center ( Site 0555), Rozzano, Milano
  - A.O. di Rilievo Nazionale e di alta Specializzazione Garibaldi ( Site 0553), Catania
  - ASST Grande Ospedale Metropolitano Niguarda ( Site 0550), Milan
  - Universita degli Studi della Campania Luigi Vanvitelli-UOC Oncoematologia ( Site 0556), Napoli
- Japan (8):
  - National Cancer Center Hospital East ( Site 0600), Kashiwa, Chiba
  - Kagawa University Hospital ( Site 0608), Kita-gun, Kagawa-ken
  - Kindai University Hospital ( Site 0607), Sayama, Osaka
  - Saitama Prefectural Cancer Center ( Site 0603), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center ( Site 0605), Sunto-gun,, Shizuoka
  - National Hospital Organization Kyushu Cancer Center ( Site 0609), Fukuoka
  - National Cancer Center Hospital ( Site 0601), Tokyo
  - Japanese Foundation for Cancer Research ( Site 0602), Tokyo
- Malaysia (4):
  - Pantai Hospital Kuala Lumpur ( Site 1303), Bangsar, Kuala Lumpur
  - Institut Kanser Negara - National Cancer Institute ( Site 1302), Putrajaya, Putrajaya
  - Beacon Hospital Sdn Bhd ( Site 1305), Petaling Jaya, Selangor
  - University Malaya Medical Centre ( Site 1301), Kuala Lumpur
- Norway (5):
  - Akershus universitetssykehus ( Site 1352), Loerenskog, Akershus
  - St Olavs Hospital ( Site 1354), Trondheim, Sor-Trondelag
  - Universitetssykehuset i Nord Norge. ( Site 1355), Tromsø, Troms
  - Helse Bergen HF - Haukeland univeritetssykehus ( Site 1353), Bergen, Vestfold
  - Oslo Universitetssykehus HF. Ulleval ( Site 1351), Oslo
- Russia (9):
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 0871), Ufa, Baskortostan, Respublika
  - SRBHI of Kirov Region Center of Oncology and medical radiology ( Site 0854), Kirov, Kirov Oblast
  - Main Military Clinical Hospital n.a. N.N.Burdenko ( Site 0870), Moscow, Moscow
  - FSBI-FRCC of Special Types Med. Care and Technologies FMBA of Russia ( Site 0851), Moscow, Moscow
  - City Hospital #40 ( Site 0853), Saint Petersburg, Sankt-Peterburg
  - Clinical Research Center of specialized types medical care-Oncology ( Site 0860), Saint Petersburg, Sankt-Peterburg
  - Tomsk National Research Medical Center of Russian Academy of Sciences ( Site 0872), Tomsk, Tomsk Oblast
  - Yaroslavl Regional SBIH Clinical Oncology Hospital ( Site 0850), Yaroslavl, Yaroslavl Oblast
  - SHBI "Leningrad Regional Clinical Oncology Dispensary n.a. L.D. Roman"-Clinical Trials Department (, Saint Petersburg
- South Africa (4):
  - Cancer Care Langenhoven Drive Oncology Centre ( Site 1504), Port Elizabeth, Eastern Cape
  - Sandton Oncology Medical Group PTY LTD ( Site 1501), Sandton, Gauteng
  - Cape Town Oncology Trials Pty Ltd ( Site 1506), Kraaifontein, Western Cape
  - Cancercare Rondebosch Oncology ( Site 1509), Rondebosch, Western Cape
- South Korea (4):
  - Asan Medical Center ( Site 0650), Songpagu, Seoul
  - Seoul National University Hospital ( Site 0653), Seoul
  - Severance Hospital ( Site 0652), Seoul
  - Samsung Medical Center ( Site 0651), Seoul
- Spain (5):
  - Hospital Universitari Vall d Hebron ( Site 0900), Barcelona
  - Hospital Sant Pau i la Santa Creu ( Site 0905), Barcelona
  - Hospital Clinico San Carlos ( Site 0902), Madrid
  - Hospital Universitario 12 de Octubre ( Site 0901), Madrid
  - Hospital Universitario Virgen Macarena ( Site 0906), Seville
- Taiwan (6):
  - Chang Gung Medical Foundation - Kaohsiung ( Site 0956), Kaohsiung City, Changhua
  - China Medical University Hospital ( Site 0953), Taichung
  - National Cheng Kung University Hospital ( Site 0955), Tainan
  - National Taiwan University Hospital ( Site 0950), Taipei
  - Taipei Veterans General Hospital ( Site 0951), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 0952), Taoyuan District
- Turkey (Türkiye) (8):
  - Baskent Universitesi Dr. Turgut Noyan Uygulama ve Arastirma Merkezi ( Site 1007), Adana
  - Acibadem Adana Hastanesi ( Site 1008), Adana
  - Gulhane Egitim ve Arastirma Hastanesi ( Site 1009), Ankara
  - Hacettepe Universitesi Tip Fakultesi ( Site 1003), Ankara
  - Ankara Sehir Hastanesi ( Site 1005), Ankara
  - Antalya Egitim ve Arastirma Hastanesi ( Site 1010), Antalya
  - Goztepe Prof.Dr. Suleyman Yalcin Sehir Hastanesi ( Site 1002), Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi ( Site 1006), Izmir
- Ukraine (4):
  - Municipal Non-Profit Enterprise City Clinical Hospital 4 of Dnipro City Council ( Site 1657), Dnipro, Dnipropetrovsk Oblast
  - MI Precarpathian Clinical Oncology Center ( Site 1654), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Ukrainian Center of Tomotherapy ( Site 1658), Kropyvnytskyi, Kirovohrad Oblast
  - Odessa Regional Clinical Hospital ( Site 1664), Odesa, Odesa Oblast
- United Kingdom (7):
  - University College London Hospitals NHS Foundation Trust ( Site 1056), London, Camden
  - Royal Marsden NHS Foundation Trust ( Site 1064), London, London, City of
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital ( Site 1052), London, London, City of
  - Royal Marsden NHS Trust ( Site 1063), Sutton, London, City of
  - University Hospital Coventry & Warwickshire ( Site 1062), Coventry, Warwickshire
  - Velindre Cancer Centre ( Site 1058), Cardiff
  - Leeds Teaching Hospitals NHS Trust ( Site 1050), Leeds

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26350&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- Favezelimab/Pembrolizumab: Participants received coformulated favezelimab/pembrolizumab (800 mg/200 mg) intravenously (IV) on Day 1, then every 3 weeks (Q3W), for up to 35 infusions.
- Standard of Care (Regorafenib or TAS-102): At the Investigator's choice, participants received 160 mg regorafenib orally daily on Days 1-12 of each 28-day cycle OR 35 mg/m^2 TAS-102 orally twice daily on Days 1-5 and Days 8-12 of each 28-day cycle.
Period: Overall Study
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Started | 221 | 220
Treated | 221 | 210
Completed | 0 | 0
Not Completed | 221 | 220
Not completed — Death | 199 | 196
Not completed — Physician Decision | 4 | 2
Not completed — Sponsor Decision | 14 | 11
Not completed — Withdrawal by Subject | 4 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102) | Total
Number analyzed (Participants) | 221 | 220 | 441
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (11.3) | 57.6 (11.4) | 58.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 81 | 164
  Male | 138 | 139 | 277
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 17 | 36
  Not Hispanic or Latino | 197 | 196 | 393
  Unknown or Not Reported | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 67 | 65 | 132
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 145 | 147 | 292
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 4 | 2 | 6
Geographic Region [Count of Participants; unit: Participants] — Randomization of participants was stratified by the geographic region of the participants (Asia Pacific or Europe, the Middle East and Africa [EMEA]/Americas).
  Participants
    Asia Pacific | 71 | 70 | 141
    EMEA/Americas | 150 | 150 | 300
Presence of Liver Metastasis [Count of Participants; unit: Participants] — Randomization of participants was stratified by the presence of liver metastasis (Yes or No).
  Participants
    Yes | 172 | 173 | 345
    No | 49 | 47 | 96
Time from Initial Diagnosis of Metastatic Disease to Randomization [Count of Participants; unit: Participants] — Randomization of participants was stratified by the time from initial diagnosis of metastatic disease to randomization (≥18 months or <18 months).
  Participants
    ≥18 months | 144 | 150 | 294
    <18 months | 77 | 70 | 147

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: Up to approximately 33 months
Population: All randomized participants were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 221 | 220
Months | 7.3 [5.8 to 8.8] | 8.5 [7.5 to 9.9]
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Superiority; p = 0.4183, Log Rank — One-sided p-value based on log-rank test stratified by geographic region (Asia Pacific; EMEA/Americas), presence of liver metastasis (Yes/No) and time from initial diagnosis of metastatic disease to randomization (>=18 months, <18 months); Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.80 to 1.20] — HR and 95% CI were based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region, presence of liver metastasis & time from initial diagnosis of metastatic disease to randomization

2. Secondary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 by BICR or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
Time Frame: Up to approximately 21 months
Population: All randomized participants were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 221 | 220
Months | 2.1 [2.1 to 2.1] | 2.6 [2.2 to 3.3]
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Superiority; p = 0.9967, Log Rank — One-sided nominal p-value based on log-rank test stratified by geographic region (Asia Pacific; EMEA/Americas), presence of liver metastasis (Yes/No) and time from initial diagnosis of metastatic disease to randomization (>=18 months, <18 months); Hazard Ratio (HR) = 1.34, 95% CI 2-sided [1.09 to 1.64] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR
Description: ORR was defined as the percentage of participants who achieved a confirmed complete response (CR: Disappearance of all target lesions) or partial response (PR: At least a 30% decrease in the sum of diameters of target lesion) per RECIST 1.1 as assessed by BICR.
Time Frame: Up to approximately 21 months
Population: All randomized participants were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 221 | 220
Percentage of Participants | 6.8 [3.8 to 10.9] | 0.9 [0.1 to 3.2]
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Superiority; p = 0.0007, Miettinen & Nurminen Method — One-sided, nominal p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in percentage = 5.9, 95% CI 2-sided [2.5 to 10.1] — Difference in percentage and 95% CI were based on the Miettinen & Nurminen method stratified by geographic region, presence of liver metastasis & time from initial diagnosis of metastatic disease to randomization

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR
Description: For participants who demonstrate confirmed CR (disappearance of all target lesions) or PR (At least a 30% decrease in the sum of diameters of target lesions), duration of response was defined as the time from the first documented evidence of CR or PR until progressive disease (PD) or death due to any cause. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions as well as an absolute increase of at least a 5 mm in the sum of diameters. The appearance of one or more new lesions was also considered PD. DOR assessments were based on blinded central imaging review with confirmation.
Time Frame: Up to approximately 21 months
Population: All randomized participants who experienced a confirmed CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 15 | 2
Months | NA [5.7 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | NA [NA to NA] — NA = Median, lower limit, and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

5. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to approximately 31 months
Population: All randomized participants who received at least one dose of study intervention were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 221 | 210
Participants | 205 | 199

6. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 28 months
Population: All randomized participants who received at least one dose of study intervention were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 221 | 210
Participants | 21 | 19

7. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score
Description: The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life (QoL; "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) is computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome.
Time Frame: Baseline and up to approximately 8 weeks
Population: All randomized participants who have received at least one dose of the study intervention and had at least one EORTC QLQ-C30 assessment data available for this outcome measure were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 217 | 205
Score on a scale | -7.11 [-9.95 to -4.26] | -4.03 [-7.05 to -1.00]
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Other; p = 0.1318, t-test, 2 sided — Two-sided p-value based on t-test; Difference in Least Square (LS) Means = -3.08, 95% CI 2-sided [-7.09 to 0.93] — Calculated using a cLDA model with PRO scores as response variable with covariates for treatment by study visit interaction & stratified by geographic region, presence of liver metastasis & time from diagnosis of metastatic disease to randomization

8. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Physical Functioning (Items 1-5) Score
Description: The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 5 questions about their physical functioning (Items 1-5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome
Time Frame: Baseline and up to approximately 8 weeks
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 217 | 205
Scores on a scale | -7.13 [-9.86 to -4.40] | -6.17 [-9.08 to -3.27]
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Other; p = 0.6370, t-test, 2 sided — Two-sided p-value based on t-test; Difference in LS Means = -0.95, 95% CI 2-sided [-4.93 to 3.02] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Appetite Loss (Item 13) Score
Description: The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire, including a single-item scale score for appetite loss (QLQ-C30 Item 13). For this item, individual responses to the question "Have you lacked appetite?" are given on a 4-point scale (1=Not at all; 4=Very much). Scores are transformed to a range from 0-100, with a lower score indicating a better outcome. The change from baseline in the EORTC QLQ-C30 appetite loss (Item 13) scale score will be presented.
Time Frame: Baseline and up to approximately 8 weeks
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 217 | 205
Score on a scale | 8.04 [3.93 to 12.15] | 4.18 [-0.16 to 8.53]
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Other; p = 0.1846, t-test, 2 sided — Two-sided p-value based on t-test; Difference in LS Means = 3.86, 95% CI 2-sided [-1.85 to 9.57] — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Change From Baseline in EORTC Quality of Life Questionnaire-Colorectal Cancer-Specific 29 Items (QLQ-CR29) Bloating (Item 37) Score
Description: The EORTC QLQ-CR29 is a health-related quality-of life (QoL) questionnaire specific for colorectal cancer, including a single-item scale score for bloating (QLQ-CR29 Item 37). For this item, individual responses to the question "Did you have a bloated feeling in your abdomen?" are given on a 4-point scale (1=Not at all; 4=Very much). Scores are transformed to a range from 0-100, with a lower score indicating a better outcome. The change from baseline in the EORTC QLQ-CR29 bloating (Item 37) scale score will be presented.
Time Frame: Baseline and up to approximately 8 weeks
Population: All randomized participants who have received at least one dose of the study intervention and had at least one EORTC QLQ-CR29 assessment data available for this outcome measure were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 217 | 205
Score on a scale | 4.33 [0.37 to 8.30] | 3.77 [-0.44 to 7.98]
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Other; p = 0.8410, t-test, 2 sided — Two-sided p-value based on t-test; Difference in LS Means = 0.56, 95% CI 2-sided [-4.96 to 6.08] — [estimate comment as in outcome 7, analysis 1]

11. Secondary Outcome: Time to Deterioration (TTD) in EORTC QLQ-C30 GHS (Item 29) and QoL (Item 30) Combined Score
Description: TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (decrease) from baseline in GHS (EORTC QLQ-C30 Item 29) & QoL combined score (EORTC QLQ-C30 Item 30). The combined score of GHS (Item 29) and QoL (Item 30) was computed by averaging raw scores of the 2 items and applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in GHS and QoL combined score, will be presented. A longer TTD indicates a better outcome.
Time Frame: Baseline and up to approximately 38 months
Population: All randomized participants who have received at least one dose of the study intervention and had EORTC QLQ-C30 assessment data available at baseline for this outcome measure were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 210 | 193
Months | NA [NA to NA] — NA = Median, lower and upper limit were not reached due to insufficient number of participants with an event. | NA [14.4 to NA] — NA = Median and upper limit were not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Other; p = 0.5094, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.64 to 1.58] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: TTD in EORTC QLQ-C30 Physical Functioning (Items 1-5) Combined Score
Description: TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (decrease) from baseline in physical functioning score (EORTC QLQ-C30 Items 1-5). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in GHS and QoL combined score, will be presented. A longer TTD indicates a better outcome.
Time Frame: Baseline and up to approximately 38 months
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 210 | 193
Months | NA [9.1 to NA] — NA = Median and upper limit were not reached due to insufficient number of participants with an event. | 20.3 [10.9 to NA] — NA = Upper limit was not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Other; p = 0.9704, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [0.98 to 2.33] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: TTD in in EORTC QLQ-C30 Appetite Loss (Item 13) Score
Description: TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (decrease) from baseline in appetite loss score (EORTC QLQ-C30 Item 13). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in physical functioning score, will be presented. A longer TTD indicates a better outcome.
Time Frame: Baseline and up to approximately 38 months
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 210 | 193
Months | NA [NA to NA] — NA = Median, lower and upper limit were not reached due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, lower and upper limit were not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Other; p = 0.9905, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.82, 95% CI 2-sided [1.11 to 2.98] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: TTD in EORTC Quality of Life Questionnaire-Colorectal Cancer-Specific 29 Items (QLQ-CR29) Bloating (Item 37) Score
Description: TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (decrease) from baseline in bloating score (QLQ-CR29 Item 37). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in appetite loss score, will be presented. A longer TTD indicates a better outcome.
Time Frame: Baseline and up to approximately 38 months
Population: All randomized participants who have received at least one dose of the study intervention and had EORTC QLQ-CR29 assessment data available at baseline for this outcome measure were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
Number analyzed (Participants) | 208 | 191
Months | NA [17.4 to NA] — NA = Median and upper limit were not reached due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, lower and upper limit were not reached due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Favezelimab/Pembrolizumab vs Standard of Care (Regorafenib or TAS-102); Test type: Other; p = 0.9853, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.86, 95% CI 2-sided [1.06 to 3.26] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to approximately 38 months
Description: Serious and Other adverse events (AEs) includes all participants who received ≥1 dose of study drug. All-Cause Mortality includes all randomized participants. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Data are reported by treatment received.
Arm/Group | Favezelimab/Pembrolizumab | Standard of Care (Regorafenib or TAS-102)
All-Cause Mortality (participants affected / at risk) | 202/221 | 203/220
Serious Adverse Events (participants affected / at risk) | 75/221 | 56/210
Other Adverse Events (participants affected / at risk) | 193/221 | 187/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Favezelimab/Pembrolizumab (N=221) | Standard of Care (Regorafenib or TAS-102) (N=210)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Addison's disease (Endocrine disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 2 (2)
Colitis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 3 (5)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (6) | 3 (3)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Anal fistula infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Favezelimab/Pembrolizumab (N=221) | Standard of Care (Regorafenib or TAS-102) (N=210)
Anaemia (Blood and lymphatic system disorders) | 33 (36) | 48 (55)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 35 (73)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 13 (21)
Hyperthyroidism (Endocrine disorders) | 26 (28) | 1 (1)
Hypothyroidism (Endocrine disorders) | 35 (36) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 20 (20) | 22 (24)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 13 (19)
Constipation (Gastrointestinal disorders) | 20 (24) | 29 (35)
Diarrhoea (Gastrointestinal disorders) | 36 (44) | 42 (65)
Nausea (Gastrointestinal disorders) | 35 (35) | 48 (66)
Vomiting (Gastrointestinal disorders) | 22 (29) | 24 (35)
Asthenia (General disorders) | 26 (27) | 21 (25)
Fatigue (General disorders) | 53 (58) | 43 (49)
Pyrexia (General disorders) | 27 (31) | 13 (18)
COVID-19 (Infections and infestations) | 15 (16) | 26 (26)
Urinary tract infection (Infections and infestations) | 9 (10) | 17 (22)
Infusion related reaction (Injury, poisoning and procedural complications) | 13 (16) | 0 (0)
Alanine aminotransferase increased (Investigations) | 23 (27) | 15 (19)
Aspartate aminotransferase increased (Investigations) | 30 (37) | 22 (25)
Blood alkaline phosphatase increased (Investigations) | 17 (17) | 13 (13)
Blood bilirubin increased (Investigations) | 13 (14) | 21 (24)
Lipase increased (Investigations) | 13 (15) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 32 (59)
Platelet count decreased (Investigations) | 2 (2) | 20 (26)
Weight decreased (Investigations) | 20 (20) | 25 (25)
White blood cell count decreased (Investigations) | 0 (0) | 21 (27)
Decreased appetite (Metabolism and nutrition disorders) | 48 (50) | 24 (26)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 17 (20) | 6 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 16 (17) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (15) | 13 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (23) | 16 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 0 (0)
Headache (Nervous system disorders) | 13 (14) | 15 (16)
Proteinuria (Renal and urinary disorders) | 13 (17) | 18 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 15 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 14 (14)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 45 (51)
Pruritus (Skin and subcutaneous tissue disorders) | 23 (25) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 18 (19) | 8 (10)
Hypertension (Vascular disorders) | 11 (12) | 28 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT05064059/Prot_SAP_000.pdf